CLINICAL TRIAL: NCT03943706
Title: Investigation of Electronic Cigarette and Cigarette Nicotine Delivery and Abuse Liability in Cigarette Smokers and Dual Users
Brief Title: E-Cigarette and Cigarette Nicotine Delivery and Abuse Liability in Cigarette Smokers and Dual Users
Status: Withdrawn | Type: Observational
Why Stopped: The investigator moved to another institution, therefore the study was never initiated.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 8841
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Tobacco Use
Keywords: e-cigarettes; JUUL brand e-cigarette; NJOY brand e-cigarette; EVOLV brand mod e-cigarette; Very Low Nicotine Cigarettes (VLNCs)
MeSH Terms: conditions — Tobacco Use; Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — During their PK (Pharmacokinetics) visits, Blood will be collected during specific time points and plasma will be extracted from the blood. Plasma will be used to analyze the levels of nicotine in it.
  Urine will be collected from female participants in order to confirm their pregnancy status. Saliva will be collected during their screening visit to analyze for cotinine levels in order to check their smoking status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exclusive cigarette smokers: Exclusive cigarette smokers must smoke at least 10 cigarettes per day for the past three months and have exhaled carbon monoxide (eCO) levels of at least 6 ppm at the screening visit.
- Dual (Electronic cigarette and cigarette smoking) users: Dual e-cigarette and cigarette users must have smoked at least 5 cigarettes per day for the last 3 months and use e-cigarettes at least 15 days per month for the last 3 months.

SUMMARY:
The FDA has shown clear interest in strategies that will reduce the public health burden of tobacco use. One proposed strategy includes banning the sale of fully nicotinized cigarettes and only allowing VLNCs (Very Low Nicotine Cigarettes) to be sold. While there are concerns regarding the unintended consequences (e.g., black market sales of fully nicotinized cigarettes) of such bans, research is needed to understand how smokers and dual users will act in the potential market. The overall aim of the current research is to understand purchasing and product choice behaviors of tobacco/nicotine users if the proposed ban were to go into effect.

DETAILED DESCRIPTION:
Tobacco use continues to be the leading cause of preventable death in the US, with the majority of deaths due to combustible tobacco use. Electronic cigarettes (e-cigarettes) may represent a nicotine delivery device that addresses cravings and nicotine withdrawal and is much less harmful compared to cigarettes, particularly if completely substituted for cigarettes. The Food and Drug Administration (FDA) recently set forth plans that include the possibility of regulating the level of nicotine in combustible cigarettes to make them non-addictive and disallowing the sale of fully nicotinized cigarettes. While studies have shown that lowering the level of nicotine in cigarettes leads to high quit rates and would likely have a positive overall public health impact, there are concerns that doing so will lead to a black market for purchasing fully nicotinized cigarettes. However, no empirical evidence currently exists regarding this possible unintended consequence of the proposed regulation and the current project aims to fill this gap. Current smokers and dual cigarette and e-cigarette users will complete three in-lab study visits. Following screening and practice with all study products, participants will complete standardized 10-puff bouts for three e-cigarettes, the VLNCs (Very Low Nicotine Cigarettes), and their usual brand cigarette. They will then complete three concurrent choice tasks. The tasks will simulate 1) the current market, in which e-cigarettes and fully nicotinized cigarettes are available, 2) the potential future market in which e-cigarettes and VLNC (Very Low Nicotine Cigarettes) are freely available and nicotinized cigarettes are banned, and 3) the potential future market in which only tobacco flavored e-cigarettes and VLNCs (Very Low Nicotine Cigarettes) are freely available and nicotinized cigarettes are banned. Understanding, in an environment where VLNCs (Very Low Nicotine Cigarettes) are the only cigarettes available, current smokers' and dual users' product choices will fill an important gap in the research and inform regulation of these products.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years old
* live within 30 miles of the research site
* interested in/willing to use an e-cigarette during study visits
* be willing and able to complete study procedures including specimen collection, survey completion, and remaining nicotine abstinent for 12 hours prior to each study visit
* speak and understand English
* willing to provide informed consent
* bring usual brand cigarettes to screener study visit.

Additional Inclusion criteria for smokers:

* smoke at least 10 cigarettes per day for the past three months,
* exhaled more than equal to 6 ppm carbon monoxide at the screener visit.

Additional Inclusion criteria for dual users:

* smoke more than equal to 5 tobacco cigarettes per day for the last 3 months,
* use e-cigarettes at least 15 days per month for the last 3 months, and
* bring e-cigarette device to screener study visit.

Exclusion Criteria:

* currently suffering from lung disease including asthma, cystic fibrosis (CF), or chronic obstructive pulmonary disease (COPD), unless it is well-controlled,
* currently pregnant or breast-feeding or have plans to become pregnant or begin breast-feeding at any point during the study,
* intoxicated at study visits (breath alcohol testing and clean urine drug screen),
* any known allergies or sensitivity to the known major constituents contained in the aerosol of the study e-cigarette devices (e.g., flavorants, vegetable glycerin, propylene glycol),
* User of zero-nicotine e-cigarettes,
* smokes mentholated cigarettes regularly,
* history of cardiac event or distress within the past 3 months.

Additional Exclusion criteria for smokers:

* have previously used any e-cigarette device (cig-a-like, pen style, mod, APV) for longer than 30 days
* use of an e-cigarette device over the past 14 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A sample of 40 current cigarette smokers (n=20) and dual e-cigarette and cigarette users (n=20) who are willing to use/try an alternative nicotine-delivery device will be recruited via advertisements/ recruitment materials (e.g., craigslist, ads on OSU, OU, and UCO campuses, OUHSC, email) and referrals. Participants will live in the Oklahoma City, OK metro area. Participants will be provided information about the study and provide initial consent for screening via an online screener.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Nicotine delivery measured by serum (blood) nicotine | 1 month
  Participants will complete one standardized puffing bout (10 puffs) with each of the three electronic cigarettes, usual brand cigarette and Very Low Nicotine Cigarettes (VLNCs). Serum nicotine will be measured throughout each standardized puffing bout. Greater levels of serum nicotine will be indicative of greater nicotine delivery.
Proportion of puffs earned and allocated to each product in three hypothetical tobacco regulatory scenarios | 1 month
  Participants will complete three computer tasks simulating hypothetical regulatory scenarios and will earn and allocate puffs to study products. A greater proportion of puffs allocated will indicate greater demand for the product in that hypothetical scenario

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Wagener, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center Oklahoma Tobacco Research Center, Oklahoma City, Oklahoma, United States